CLINICAL TRIAL: NCT06532084
Title: Randomized Trial of Sorafenib Prophylaxis After Allogeneic Hematopoietic Stem Cell Transplantation With Post-transplantation Bendamustine and Cyclophosphamide
Brief Title: Sorafenib Relapase Prophylaxis After HCT With PTBCy Regimen
Acronym: SoraGVL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: St. Petersburg State Pavlov Medical University (Other)
Responsible Party: Principal Investigator, Ivan S Moiseev, Vice-director of RM Gorbacheva Research Institute, St. Petersburg State Pavlov Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19/24-n
Record Dates: First submitted 2024-07-29; First posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Acute Myeloid Leukemia, in Relapse; Myelodysplastic Syndromes; Chronic Myeloid Leukemia; Myeloproliferative Neoplasm
Keywords: post-transplantation cyclophosphamide; post-transplantation bendamustine; acute myeloid leukemia; myelodysplastic syndrome; refractory; sorafenib
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Myeloproliferative Disorders | interventions — Sorafenib

STUDY DESIGN:
Intervention Model Description: In total 88 patients will be included in the study. After inclusion into the study patients will be randomized in 1:1 proportion in two arms (44 patients per arm): treatment with sorafenib or observation. Patients will be followed up for two years. The strata is a type of donor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sorafenib prophylaxis (Experimental): Sorafenib 200 mg bid for 168 days starting before day+100 after HCT
  Interventions: Drug: Sorafenib
- Observation (No Intervention): Usual care

INTERVENTIONS:
Drug: Sorafenib — Sorafenib 200 mg bid for 168 days starting in the time fram between engraftment with neutrophils > 1.0 x 10^9/L, white blood cells> 1.5 x 10^9/L, platelets> 1.5 x 10^9/L and day+100 after allogeneic hematopoietic cell trnaplantation
  Arms: Sorafenib prophylaxis

SUMMARY:
This is a single-center randomized open-label phase II clinical trial to compare relapse prophylaxis with sorafenib and observation after graft-versus-host disease prophylaxis with post-transplantation bendamustine and cyclophosphamide in high-risk myeloid malignancies. This is an intention to treat study, where randomization is performed at first documentation of CR after engraftment.

DETAILED DESCRIPTION:
Allogeneic hematopoietic stem cell transplantation (HCT) results steadily improve due to reduction of NRM. Standard risk patients now have the risk of HCT below 10% after matched donor transplantation. Nonetheless, there is limited improvement in CIR over time. Especially novel strategies to reduce relapse are needed for high-risk myeloid malignancies where standard HCT approaches result in relatively unfavorable outcomes. Among high-risk malignancies are refractory AML without hematological remission for HCT. In this group EFS rarely exceeds 15%. Some improvement in refractory AML was reported with intensified sequential conditioning regimens, but there use is limited to young and fit patients who comprise only around 20-30% of all refractory AML population. Also it was demonstrated that AML patients beyond CR2 have significantly worse prognosis than CR1 and CR2 patients. It is reported that long-term EFS in this group of patients is around 30%. The next adverse group of HCT recipients are patients with high-risk somatic mutations. It is reported in several studies that EFS in tp53-mutant AML even allografted in CR is 0%. Another adverse mutation is ASXL1, where also 0-10% EFS was demonstrated in large cohorts of patients. For therapy related myeloid malignancies it was also demonstrated that the CIR is higher and this group patients have even in CR have 30% EFS. Complex karyotype and monosomal karytope, involvement of chromosome 3 with EVI1 gene, which are common in this patients group, further exacerbate prognosis. Very high risk MDS was also reported to have dismal prognosis after allogeneic HCT. All these adverse groups were included in the study.

PTBCy GVHD prophylaxis provides augmented GVL and better disease control in high-risk myeloid malignancies, but GVL effect fades over time. While median relapse rate is significantly prolonged to 8 months against the previously reported in the literature 2-3 months, the relapse rate with long term follow up remains high. Thus this longer time to relapse gives enough time to initiate sorafenib prophylaxis which was shown to be one of the most promising agents for relapse prophylaxis. Given its immune modulatory properties the study hypothesis is that sorafenib with PTBCy GVHD prohylaxis will further augment GVL and facilitate better disease control.

ELIGIBILITY:
Inclusion Criteria:

* Patients must undergo allogeneic hematopoietic stem cell transplantation with post-transplantation bendamustine AND cyclophosphamide from any donor.
* Patients must have high-risk myeloid malignancy as an indication for transplantation defined as:

  * acute myeloid leukemia not in hematological remission prior to transplantation,
  * ≥ 3 remission of acute myeloid leukemia,
  * any myeloid malignancy with bi-allelic tp53 mutation,
  * any myeloid malignancy with complex karyotype,
  * therapy-related myeloid malignancy not in MRD-negative response
  * myelodysplastic syndrome with very high IPSS-R risk
  * any myeloid malignancy with monosomal or t(3;3) karyotype,
  * any myeloid malignancy with ASXL1, bi-allelic tp53 or RUNX1 mutation, EVI1 overexpression
  * MDS/NPM unclassified not in hematologic remission.
* Documented hematological remission in the bone marrow at the time of inclusion post-engraftment, measurable residual disease is allowed
* First 100 days after allogeneic hematopoietic stem cell transplantation

Exclusion Criteria:

* successfully treated relapse between transplantation and enrollment
* use of any other planned method for prophylaxis of relapse besides sorafenib
* donor lymphocyte infusion prior to randomization
* Second malignancy not in complete remission within 6 months prior to randomization
* Moderate or severe cardiac disease: ejection fraction <50%, unstable angina, stable angina NYHA class III or IV, chronic heart failure NYHA class III or IV, Lawn grade V arrhythmia, myocardial infarction within 3 months before inclusion
* Stroke within 3 months of inclusion, unless related to the underlying malignancy
* Severe decrease in pulmonary function: FEV1 <50% or DLCO<50% of predicted or respiratory distress or need for oxygen support;
* Severe organ dysfunction: AST or ALT >10 upper normal limits, bilirubin >2 upper normal limits, creatinine >2 upper normal limits
* Creatinine clearance < 30 mL/min
* Uncontrolled bacterial or fungal infection at the time of enrollment defined by CRP> 70 mg/L
* Requirement for vasopressor support at the time of enrollment
* Requirement for positive-pressure oxygen at the time of enrollment
* Karnofsky index <30%
* Pregnancy
* Somatic or psychiatric disorder making the patient unable to sign informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2024-05-22 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Event-free survival | 2 years
  Kaplan-Meier estimate of either relapse or secondary graft failure or death from all causes

SECONDARY OUTCOMES:
Overall survival | 2 years
  Kaplan-Meier estimate of death from all causes
Cumulative incidence of primary and secondary graft failure | 365 days
  Cumulative secondary graft failure, competing risk is death and relapse
Incidence of HCT-associated adverse events | 180 days
  Toxicity assessment is based on presence of NCI CTC AE 5.0 event grades 3-5. Veno-occlusive disease incidence and severity assessment is based on EBMT criteria 2020. Transplant-associated microangiopathy incidence assessment is based on Harmonization criteria. All toxicity measurements will be aggregated as severity scores.
Infectious complications, including analysis of severe bacterial, fungal and viral infections incidence | 180 days
  proportion of patients, requiring systemic treatment for bacterial, viral and fungal diseases
Cumulative incidence of acute GVHD grade II-IV | Cumulative incidence of patients with acute GVHD II-IV grade, competing risk is death, relapse and graft failure
  125 days
Cumulative incidence of moderate and severe chronic GVHD | 2 years
  Cumulative incidence of patients with moderate and severe chronic GVHD according to NIH 2015 criteria, competing risk is death, relapse and primary graft failure
Non-relapse mortality analysis | 2 years
  Cumulative incidence of patients with mortality without hematological relapse of malignancy
GVHD-relapse-free survival analysis | 2 years
  Kaplan-Meier estimate of death, acute GVHD grade III-IV, severe chronic GVHD or relapse
Cumulative incidence of relapse | 2 years
  Cumulative incidence of patients with relapse, competing risk is non-relapse mortality

CONTACTS AND LOCATIONS:
Locations (1):
- RM Gorbacheva Research Institute, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: Yes
Upon written study proposal according to Pavlov University LEC SOPs.
Supporting Information: Study Protocol
URL: https://cloud.mail.ru/public/pWy9/SHFTSkm6Y